CLINICAL TRIAL: NCT02424175
Title: Fecal Microbiota Transplantation for the Treatment of Primary Sclerosing Cholangitis.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joshua Korzenik, Director, Crohn's and Colitis Center, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P002475
Record Dates: First submitted 2015-04-18; First posted 2015-04-22 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-08

CONDITIONS: Sclerosing Cholangitis
Keywords: Fecal Transplant; Primary Sclerosing Cholangitis; Fecal Microbiota Transplantation
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with PSC (Experimental): This is an open label study. All patients enrolled will receive a fecal microbiota transplantation.
  Interventions: Biological: Fecal Microbiota Transplantation

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation

SUMMARY:
This is an open-label single-arm pilot study to measure the safety, microbiological and clinical impacts of Fecal Microbiota Transplantation (FMT) in patients with Primary Sclerosing Cholangitis (PSC). The investigators will prospectively enroll 10 PSC patients Stage 1 and 2 who also have concurrent inflammatory bowel disease Donor Stool from one healthy donor will be obtained from OpenBiome. OpenBiome is a nonprofit 501(c)(3) organization that provides hospitals with screened, filtered, and frozen material ready for clinical use

DETAILED DESCRIPTION:
Background and Significance:

Primary sclerosing cholangitis (PSC) is a progressive, chronic cholestatic liver disease characterized by inflammatory and fibrotic destruction of the intrahepatic and/or extrahepatic bile ducts. PSC will progress to biliary cirrhosis, portal hypertension and liver failure (1) . It is a common indication for liver transplantation. In up to 90% of patients, ulcerative colitis or Crohn's disease will also be present (2) . Medications used for the treatment of ulcerative colitis such as sulfasalazine, corticosteroids and azathioprine or 6-mercaptopurine have not been effective in reducing inflammation or bringing about remission in PSC (3) . A number of studies of other anti-inflammatory agents have failed to demonstrate any benefit. In standard dosing, ursodeoxycholic acid (UDCA) may be of benefit in delaying the progression of disease, although a recent study showed that high dose UDCA was not only ineffective, it may also be harmful (4) . Currently there is no medical therapy that has been shown to be effective in PSC and no therapy has won FDA approval for this indication.

It has been postulated that bacterial components may stimulate an aberrant immune response resulting in the perpetuation of the biliary inflammation seen in PSC. Bacteria gain access to the liver and biliary tree through translocation across an abnormal and inflamed intestinal mucosa into the portal venous system (5) . Studies have shown an increased risk of portal venous bacteremia in patients with PSC. Animal models have demonstrated that enteric dysbiosis can lead to hepatobiliary inflammation with various features of PSC (6) . The pathways through which bacteria might then induce the pathology characteristic of PSC are speculative.

Bacteria might cause direct injury through colonization, though studies have not identified any particular pathogen or a consistent set of bacteria. Another potential pathway may be that a certain set of bacteria generate secondary bile acids, such as deoxycholic acid and lithocholic acid, which are injurious to the biliary system (7) . We recently found an altered serum bile acid composition in patients with PSC compared to non-cholestatic controls. Treatment with UDCA in PSC patients decreases the concentration of the toxic primary bile acid chenodeoxycholic acid but also increased the toxic secondary bile acid lithocholic acid (Abstract DDW 2014). Alteration of the gut microbiota may minimize or eliminate this injury.

There is limited experience in the use of antibiotics in treating PSC. Metronidazole has been shown to result in improvement in liver function tests (8) . Oral vancomycin has also been advanced as a potentially promising therapy (9) . An initial report of three pediatric patients and a subsequent small, uncontrolled series of oral vancomycin in 14 children showed improvement in liver tests and symptoms (10, 11) . We recently completed a study of oral vancomycin was given to 10 adults with PSC found mild improvement in serum alkaline phosphatase levels (Abstract DDW 2011).

Fecal Biotherapy (FBT) also known as fecal transplantation or fecal microbiota transplant-involves the transfer of a donor's fecal flora (bacteria) to a recipient's colon. It has become widely accepted as the standard of care for recurrent Clostridium difficile 3 infection, with a cumulative cure rate of >90% and minimal adverse events (12) . In C. diff infection, prior exposure to antibiotics diminishes the normal colonic flora, allowing C. diff organism to proliferate and release toxin (13) . This bacterial environment is similar to the major shifts in microbial diversity seen in patients with IBD. Interestingly, when patients with IBD receive FBT for C. diff. infections, their outcomes are excellent, reinforcing the notion that the enteric flora have a strong influence in the enteric immune system (14) . We currently have a robust FMT clinical program for recurrent and refractory c.difficle infections with a cure rate > 90%. We have also recently participated in an open label clinical trial for the use of FMT in crohn's disease.

We hypothesize that for patients with PSC, fecal microbiota transplantation will correct a dysbiosis that has led to hepatobiliary inflammation leading to improvement in LFTs and slow progression to cirrhosis.

Specific Aims:

Specific Aim 1: Determine the impact of fecal microbiota transplantation on the intestinal microbiome of patients with primary sclerosis cholangitis with and without inflammatory bowel disease via 16s ribosomal RNA sequencing comparing delivery modalities (colonoscopy and capsules).

Hypothesis: Fecal microbiota transplantation will result in a sustained repopulation of the patient's microbiome that corresponds to the bacteria from the donor stool.

Specific Aim 2: Assess for clinical response in patients with PSC receiving FMT comparing delivery modalities (colonoscopy and capsules).

Hypothesis: Fecal microbiota transplantation will lead to a 50% reduction in liver biochemistries in patients with PSC.

Specific Aim 3: Assess bile salt metabolomics as a therapeutic biomarker for clinical response to fecal microbiota transplantation.

Hypothesis: A decrease in the production of toxic secondary bile acids (lithocholic and deoxycholic acid) will correlate with clinical response to fecal microbiota therapy

Primary Physiological Endpoint:

12

1. Recipient's fecal microbial diversity at 12 weeks after FMT, when compared to baseline using 16s ribosomal RNA.

Primary Clinical Endpoint

1. The primary study end point is them mean change serum liver biochemistries after 3 months of treatment as compared with baseline. Treatment success was defined as an improvement in serum alkaline phosphatase, total bilirubin, alanine aminotransferase (ALT), or aspartate aminotransferase (AST) by 50 % or greater.

Secondary Endpoints Metabolomics: Bile salt profiles of the samples and associated community structure of the fecal microbiome will be assessed as a measure of the interplay between host and gut microbiota. Stool and Serum will be analyzed using the metabolomics platform at the Broad Institute, targeting bile acids. Samples will be sent to the Broad Institute where we will use liquid chromatography tandem mass spectrometry (LC-MS) to measure endogenous bile salts and their metabolite levels in fecal supernatant. Water soluble metabolites will be extracted from feces as described by Saric et al while lipids will be extracted from lypophilized samples using isopropanol. Water soluble metabolites will be measured using ion pairing chromatography and hydrophilic interaction chromatography methods, and lipids and bile acids will be measured using C4 and C18 reversed phase chromatography methods. MultiQuant software (AB SCIEX) will be used for automated peak integration and manual review of peak quality prior to statistical analyses. The GenePattern (Broad Institute) and IPA (Ingenuity Systems) software will be used to analyze and visualize results.

Clinical Endpoints:

1. Mean change in Harvey Bradshaw Index (HBI) and PBC 40 score between week 0 and week 1, 4, 8, and 12. Percentage of patients in clinical remission (those with an HBI score at week 12 <5)
2. Mean change in Mayo Risk Score at week 12 compared to baseline. The Mayo Risk Score (MRS) for PSC is calculated based using the following formula: risk = (0.0295 * (age in years)) + (0.5373 * LN(total bilirubin in mg/dL)) - (0.8389 * (serum albumin in g/dL)) + (0.5380 * LN(AST in IU/L) + (1.2426 * (points for variceal bleeding)) If your Mayo Risk Score is less than or equal to 0 then you are in the "low" risk group. If your Mayo Risk Score is greater than 0 but less than 2 then you are in the "intermediate" risk group. If your Mayo Risk Score is greater than 2 then you are in the "high" risk group.

Safety Endpoints: Number and nature of adverse events at week 1, 4, 8, 12 and 24

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Confirmed diagnosis of PSC (with a concurrent diagnosis of inflammatory bowel disease) characterized by a cholestatic liver condition of greater than 6 months duration with confirmatory cholangiographic findings, as well as an elevation of the serum alkaline phosphatase of greater than 1.5 times the upper limit of normal.

Exclusion Criteria:

1. Decompensated liver disease
2. Patients who were pregnant or breastfeeding
3. Use of concomitant immune modulators including methotrexate, mycophenolate mofetil, tacrolimus, cyclosporine, thalidomide, Interleukin-10, or Interleukin-11 within 4 weeks prior to receiving the FMT
4. Patients who are unable to give informed consent
5. Patients who are unable or unwilling to undergo colonoscopy with moderate sedation (>ASA class II)
6. Patients who have previously undergone FMT Patients who have a confirmed malignancy or cancer
7. Patients who are immunocompromised
8. Treatment within last 8 weeks with infliximab, adalimumab, certolizumab, natalizumab, vedolizumab or thalidomide
9. Antibiotic use within 2-months of start date
10. Participation in a clinical trial in the preceding 30 days or simultaneously during this trial
11. Probiotic use within 30 days of start date
12. Congenital or acquired immunodeficiencies
13. Other comorbidities including:Diabetes mellitus, cancer, systemic lupus, must be able to tolerate conscious sedation with colonoscopy
14. Chronic kidney disease as defined by a GFR <60mL/min/1.73m2 44
15. History of rheumatic heart disease, endocarditis, or valvular disease due to risk of bacteremia from colonoscopy
16. Steroid dose >20mg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2018-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Korzenik, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study lasted from February 2016 until June 2017. 10 total patients were recruited through the Brigham and Women's Hospital Gastroenterology clinic and through referrals from other Gastroenterologists.
Pre-assignment Details: A wash out period was included for patients. All subjects should not have used antibiotics within 2 months of start date or receive treatment of infliximab, adalimumab, certolizumab, natalizumab, vedolizumab or thalidomide within the past 8 weeks. They are also screened for various infectious risks such as HIV or Hepatitis.
Groups:
- Patients With PSC: This is an open label study. All patients enrolled will receive a fecal microbiota transplantation.
  Fecal Microbiota Transplantation
Period: Overall Study
Arm/Group | Patients With PSC
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With PSC
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 41.1 [23 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Alkaline phosphatase [Mean (Full Range); unit: U/L] | 489 [111 to 1045]
Alanine Aminotransferase [Mean (Full Range); unit: U/L] | 150.7 [74 to 297]
Aspartate Aminotransferase [Mean (Full Range); unit: U/L] | 114.4 [60 to 270]

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event Frequency
Description: Number of patients with reporting adverse events irregardless of severity
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With PSC
Number analyzed (Participants) | 10
Participants | 8

2. Primary Outcome: Comparison of Alkaline Phosphatase Pre and Post Transplant
Description: The primary clinical study end point is the number of patients that achieve a 50% or more decrease serum alkaline phosphatase
Time Frame: Baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With PSC
Number analyzed (Participants) | 10
Participants | 3

3. Secondary Outcome: Microbiome
Description: Number of patients that experienced changes in the microbiome post FMT. Measured as similarity to the donor microbiome post FMT compared to their baseline sample
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With PSC
Number analyzed (Participants) | 10
Participants | 8

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 2 years from June 2016 through May 2018
Arm/Group | Patients With PSC
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With PSC (N=10)
Sinusitis (Infections and infestations) | 1 (1) — Patient had an infection that caused sinusitis and went to the ER to be treated.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With PSC (N=10)
Fever (Gastrointestinal disorders) | 2 (3)
diarrhea (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Itchiness (Skin and subcutaneous tissue disorders) | 3 (3)
MIgraine (Nervous system disorders) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1)
Polyp (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT02424175/Prot_SAP_000.pdf